CLINICAL TRIAL: NCT06296251
Title: A Randomized, Double-Blind, Placebo-Controlled, Three-Arm Parallel Study to Investigate the Effects of a Dietary Supplement Containing N-trans-Caffeoyltyramine (NCT) and N-trans-Feruloyltyramine (NFT) on Body Fat Composition
Brief Title: Dietary Supplementation on Body Fat Composition
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brightseed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BIO-2313
Record Dates: First submitted 2024-02-29; First posted 2024-03-06 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Dyslipidemias; Pre-diabetes
MeSH Terms: conditions — Dyslipidemias; Glucose Intolerance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo treatment (Placebo Comparator): Placebo treatment (Microcrystaline cellulose): 1 capsule/day
  Interventions: Other: Placebo treatment
- Active low dose of plant derived phenolics (Active Comparator): Active low dose of plant derived phenolics via 1 capsule/day
  Interventions: Dietary Supplement: Plant derived phenolics
- Active high dose of plant derived phenolics (Active Comparator): Active high dose of plant derived phenolics via 1 capsule/day
  Interventions: Dietary Supplement: Plant derived phenolics

INTERVENTIONS:
Other: Placebo treatment — Microcrystaline cellulose (MCC)
  Arms: Placebo treatment
Dietary Supplement: Plant derived phenolics — Dietary supplement containing plant derived phenolics
  Arms: Active high dose of plant derived phenolics; Active low dose of plant derived phenolics

SUMMARY:
The purpose of the current study is to examine the effects of a dietary supplement containing plant derived phenolics at two different dose levels in otherwise generally healthy adults with risk factors (high BMI at dyslipidemia and/or pre-diabetes) for body fat composition. The primary hypothesis is that supplementation with plant derived phenolics will decrease body fat composition compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, ≥18 years of age at visit 1 (week -1).
2. Body mass index (BMI) of ≥28.0 kg/m2 to <35.0 kg/m2 at visit 1 (week -1).
3. At least one of the following comorbidities based on blood draws at visit 1:

   * Dyslipidemia (any of the following)

     * Total-C ≥200 mg/dL
     * LDL-C ≥130 mg/dL
     * HDL-C ≤40 mg/dL
     * Triglycerides ≥150 mg/dL
   * Pre-diabetes o HbA1c ≥5.7 to ≤6.4% Stable use of medications allowed, where stable use is defined as the same dose for at least 90 d prior to visit1.
4. Non-user or former user (cessation ≥12 months) of tobacco or nicotine products (e.g., cigarette smoking, vaping, chewing tobacco) with no plans to begin use during the study period.
5. Willing to maintain a stable intake of current dietary supplements and medications not specifically listed as exclusionary or deemed to interfere with study outcomes throughout study duration.
6. Willing to adhere to all study procedures and signs forms providing informed consent to participate in the study and authorization to release relevant protected health information to the Clinical Investigator.

Exclusion Criteria:

1. Weight loss or gain ≥4.5 kg within 90 days of visit 1.
2. Use of weight loss medications within 90 days of visit 1
3. History of gastrointestinal surgery (e.g., bariatric surgery) or cosmetic procedures (e.g., liposuction) for weight/fat reducing purposes.
4. Use of dietary supplements or related products that, in the judgment of the Investigator, are likely to markedly affect weight loss or appetite within 30 days of visit 1.
5. History of extreme dietary habits (e.g., Atkins diet, etc.), as judged by the Investigator.
6. History of an eating disorder (e.g., anorexia nervosa, bulimia nervosa, or binge eating) diagnosed by a health professional.
7. Current medical diagnosis of type 1 or type 2 diabetes mellitus.
8. HbA1c ≥48 mmol/mol (6.5%) as measured at visit 1.
9. History of a chronic gastrointestinal disorder, such as peptic ulcer disease or malabsorption syndrome (mild lactose intolerance or gastroesophageal reflux diseases are acceptable).
10. History of liver disease with exception of non-alcoholic fatty livery disease (NAFLD).
11. Unstable use of medications for mental or emotional disorders, where stable use is defined as the same dose for ≥90 days prior to visit 1.
12. Uncontrolled stage 2 hypertension (systolic blood pressure ≥140 mm Hg or diastolic blood pressure ≥90 mm Hg) as defined by the blood pressure measured at visit 1. Participants with hypertension on a stable dose of medication may be allowed in the study per Investigator's discretion. Stable dose is defined as same dose for >90 days.
13. Habitual use (i.e., daily) of marijuana and hemp products including CBD products within 30 days of visit 1.
14. History or presence of cancer (including any malignant GI polyps) within 2 years of visit 1, except for non-melanoma skin cancer.
15. Unstable use of thyroid hormone replacement medication, where stable use is defined as the same dose for ≥90 days prior to visit 1.
16. Known intolerance or sensitivity to any ingredients in the study products.
17. Exposure to any non-registered drug product within 4 weeks prior to visit 1.
18. Signs or symptoms of an active infection of clinical relevance* within 5 days of visit 1. The visit may be rescheduled such that all signs and symptoms have resolved (at the discretion of the Clinical Investigator) at least 5 days prior to visit 1.
19. Female who is pregnant, planning to be pregnant during the study period, lactating, or is of childbearing potential and is unwilling to commit to the use of a medically approved form of contraception throughout the study period. The method of contraception must be recorded in the source document.
20. Recent history (within 12 months of visit 1) of alcohol or substance abuse. Alcohol abuse is defined as >14 drinks per week (1 drink = 12 oz. beer, 5 oz. wine, or 1½ oz. distilled spirits).
21. Any condition the Investigator believes would interfere with his or her ability to provide informed consent, comply with the study protocol, or which might confound the interpretation of the study results or put the person at undue risk. *If an infection occurs during the study period, test visits will be rescheduled until signs and symptoms have resolved (at the discretion of the Clinical Investigator) at least 5 days prior to the scheduled study visits.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-04-18 (Actual); Primary Completion 2024-12-27 (Estimated); Study Completion 2025-02-27 (Estimated)

PRIMARY OUTCOMES:
Body fat mass | 0, 12, 24 weeks
  Body fat mass (kg) change by the DEXA scan.

SECONDARY OUTCOMES:
Body composition | 0, 12, 24 weeks
  Measured by the DEXA scan:
  o Percent fat mass (%), expressed as a percentage of the total body mass
Android fat mass | 0, 12, 24 weeks
  Measured by the DEXA scan:
  o Android fat mass (kg)
Gynoid fat mass | 0, 12, 24 weeks
  Measured by the DEXA scan:
  o Gynoid fat mass (kg)
Abdominal visceral fat mass | 0, 12, 24 weeks
  Measured by the DEXA scan:
  o Abdominal visceral fat mass (g)
Abdominal circumference | 0, 12, 24 weeks
  measured by the 3D body scan:
  o Waist (abdominal) circumference (cm)
Hip circumference | 0, 12, 24 weeks
  measured by the 3D body scan:
  o Hip circumference (cm)
Chest circumference | 0, 12, 24 weeks
  measured by the 3D body scan:
  o Chest circumference (cm)
Upper thigh circumference | 0, 12, 24 weeks
  measured by the 3D body scan:
  o Upper thigh (average of left and right thighs) circumference (cm)
Upper arm circumference | 0, 12, 24 weeks
  measured by the 3D body scan:
  o Upper arm bicep (average of left and right arms) circumference (cm)
Waist to hip ratio | 0, 12, 24 weeks
  measured by the 3D body scan:
  o Waist (abdominal) to hip ratio
Fasting glucose | 0, 12, 24 weeks
  Fasting glucose through blood
Fasting insulin | 0, 12, 24 weeks
  Fasting insulin through blood
HbA1c | 0, 12, 24 weeks
  HbA1c through blood
FGF21 | 0, 24 weeks
  FGF21 through blood
Systolic blood pressure | 0, 4, 8,12, 24 weeks
  Systolic blood pressure (mmHg)
Diastolic blood pressure | 0, 4, 8,12, 24 weeks
  Diastolic blood pressure (mmHg)
Total-Cholesterol | 0, 12, 24 weeks
  Total-C through blood
HDL-C | 0, 12, 24 weeks
  HDL-C through blood
LDL-C | 0, 12, 24 weeks
  LDL-C through blood
VLDL-C | 0, 12, 24 weeks
  VLDL-C through blood
non-HDL-C | 0, 12, 24 weeks
  non-HDL-C through blood
Triglycerides | 0, 12, 24 weeks
  Triglycerides through blood
Body Weight | 0, 4, 8, 12, 16, 20, and 24 weeks
  Change in body weight from week 0 to each measured follow-up visit
Physical functioning | 0, 12, 24 weeks
  Physical functioning via 36-Item Short Form Health Survey (SF-36) questionnaire. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Bodily pain | 0, 12, 24 weeks
  Bodily pain via 36-Item Short Form Health Survey (SF-36) questionnaire. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Role limitations due to physical health | 0, 12, 24 weeks
  Role limitations due to physical health via 36-Item Short Form Health Survey (SF-36) questionnaire. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Role limitation due to personal or emotional problems | 0, 12, 24 weeks
  Role limitation due to personal or emotional problems via 36-Item Short Form Health Survey (SF-36) questionnaire. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Emotional well-being | 0, 12, 24 weeks
  Emotional well-being via 36-Item Short Form Health Survey (SF-36) questionnaire. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Social functioning | 0, 12, 24 weeks
  Social functioning via 36-Item Short Form Health Survey (SF-36) questionnaire. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Energy/Fatigue | 0, 12, 24 weeks
  Energy/Fatigue via 36-Item Short Form Health Survey (SF-36) questionnaire. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
General health perceptions | 0, 12, 24 weeks
  General health perceptions via 36-Item Short Form Health Survey (SF-36) questionnaire. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Total kcals | 0, 12, 24 weeks
  Total kcals via FFQ dietary intake parameters
Total fat | 0, 12, 24 weeks
  Total fat via FFQ dietary intake parameters
Total protein | 0, 12, 24 weeks
  Total protein via FFQ dietary intake parameters
Total carbohydrates | 0, 12, 24 weeks
  Total carbohydrates via FFQ dietary intake parameters
Fiber | 0, 12, 24 weeks
  Fiber via FFQ dietary intake parameters
Healthy Eating Index (HEI) score | 0, 12, 24 weeks
  Healthy Eating Index (HEI) score via Food Frequency Questionnaire (FFQ) dietary intake parameters. The scores range from 0 to 100. An ideal overall HEI score of 100 reflects that the set of foods aligns with key dietary recommendations and dietary patterns published in the Dietary Guidelines.
ALT | 0, 12, 24 weeks
  Changes in the chemistry profile for safety parameters
AST | 0, 12, 24 weeks
  Changes in the chemistry profile for safety parameters

CONTACTS AND LOCATIONS:
Locations (1):
- Biofortis Research, Addison, Illinois, United States